CLINICAL TRIAL: NCT00773591
Title: Effect of NT 201 (Botulinum Neurotoxin Type A Free of Complexing Proteins) on Sleep-related Breathing Disorders (Snoring Study)
Brief Title: Effect of NT 201 (Botulinum Neurotoxin Type A Free of Complexing Proteins) on Sleep-related Breathing Disorders
Acronym: Snoring
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The BfArM (CA)approved the trial in Nov 2008. However, the responsible EC refused approval in March 2009.
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Nicole Albala, Study Manager, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201 SB_2001
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Sleep-Disordered Breathing
Keywords: Sleep-related breathing disorders; Snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Typ A (Active Comparator)
  Interventions: Drug: NT 201, a Botulinum neurotoxin type A, free of complexing proteins
- Placebo (Placebo Comparator)
  Interventions: Drug: NT 201, a Botulinum neurotoxin type A, free of complexing proteins

INTERVENTIONS:
Drug: NT 201, a Botulinum neurotoxin type A, free of complexing proteins — NT 201: Solution for injection, one dose of 5 U will be administered. Route Injection into the soft palate 1 cm dorsal to the junction with the hard palate and 1 cm medial to the alveolar ridge.
  Placebo: Solution for injection, Dose n.a.; identical injected volume as active study medication. Route Injection into the soft palate 1 cm dorsal to the junction with the hard palate and 1 cm medial to the alveolar ridge.

SUMMARY:
This proof-of-concept study is to assess the potential benefit of botulinum toxin for patients with sleep-related breathing disorders.

DETAILED DESCRIPTION:
Mono-center, double-blind, 1:1 randomized, placebo-controlled trial 18 treated patients, 9 patients per group.

Patients will be randomly assigned to treatment with NT 201 or placebo in a ratio of 1:1. In addition, within each treatment group patients will be randomly assigned to injection into the left or right soft palate.

Primary variable:

Comparison of the ratio of snoring time over sleeping time (Snoring Index). Other secondary variables will be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients of at least 18 years of age.
2. Patient who understand the nature of the study and provide written informed consent prior to protocol-specific procedures.
3. Patients suffering from sleep-related breathing disorders for at least 3 months prior to study start and seeking help for their snoring.
4. Non-REM RDI ≤ 25/h (according to Medicare Criteria) at baseline PSG.
5. AHI ≤ 10/h at baseline PSG.
6. Snoring Index ≥ 15 at baseline PSG.

Exclusion Criteria:

1. Patients with known hypersensitivity to:

   * botulinum neurotoxin type;
   * any of the excipients (human albumin, sucrose).
2. Patients with upper respiratory tract pathology as assessed by an ear, nose, and throat [ENT] specialist.
3. Patients with generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert-Eaton syndrome).
4. Patients with bleeding disorders of any type and/or receiving anticoagulant therapy.
5. Patients with a profound sleep disorder (pathological number and duration of episodes of hypopnea and apnea), upper airway resistance syndrome [UARS], or obstructive sleep apnea syndrome [OSAS].
6. Obese patients (BMI ≥ 30).
7. Presence of concomitant diseases:

   * severe or unstable cardiovascular (e.g. severe angina pectoris, post myocardial infarction and ventricular extra systoles), pulmonary, or endocrine disease; clinically relevant renal or hepatic disease or dysfunction; hematological disorder; any other clinically relevant medical condition that could increase the risk to the study participant;
   * malignant disease of any kind during the previous 5 years except for successfully treated skin (basal or squamous cell) cancer;
   * amyotrophic lateral sclerosis or other diseases which result in peripheral neuromuscular dysfunction;
   * risk of developing an angle closure glaucoma;
   * alcohol, drug, or medication abuse within the past year;
   * severe psychiatric or neurological disorders;
   * acute infections of the pharynx.
8. Patients likely to need concomitant medication as follows:

   * 4-aminochinolines;
   * aminoglycosides or spectinomycin, or other medical products interfering with neuromuscular transmission, e.g. tubocurarine-type muscle relaxants;
   * daily psychotropic medication;
   * regular intake or onset of hypnotics, e.g. benzodiazepines, chloralhydrate and combinations, barbiturates (except of mild phytotherapeutics, e.g. valerian, hop and combinations);
   * anti-snoring products during the course of the study such as foams, dental devices.
9. Pregnant or nursing women, or women of childbearing potential who are not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, unless they are surgically sterilized/ hysterectomized.
10. Participation in a clinical study within the last 30 days prior to the start of the study.
11. Patients who are employees, relative or spouse of the investigator, of other staff of the investigational site or the sponsor or the CRO.
12. Any donation of germ cells, blood, organs, or bone marrow during the course of the study.
13. Patients who are expected to be non-compliant and/or not cooperative.
14. Patients who are not contractually capable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of the ratio of snoring time over sleeping time (Snoring Index) | Snoring Index measured from baseline to follow-up visit and to V3.

SECONDARY OUTCOMES:
Change in ventilation (oral/nasal flow) from V0 to V2 and from V0 to V3 including: → Peakflow Vmax → Tidal volume (Vt) | Change in several Secondary variables from baseline over time